CLINICAL TRIAL: NCT06678152
Title: Investigation of Nicotine in Umbilical Cord Tissue: Immunohistochemical and Biochemical Analysis of Cancer Stem Cell Markers
Brief Title: Nicotine's Effect on Cancer Stem Cell Markers in Human Umbilical Cord Tissue
Status: Completed | Type: Observational
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Other Study IDs: MCBU_ Nicotin_cancer
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Umbilical Cord Issue; Nicotine Addiction; Pregnancy Related; Cancer
Keywords: umblical cord; nicotine addiction; Cd44; Cd34; Cd90; ALDH
MeSH Terms: conditions — Tobacco Use Disorder; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — umblical cord tissues and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1:: smokers
- Group 2:: nonsmokers

SUMMARY:
The umbilical cord is generally an organ that clinicians and pathologists do not pay sufficient attention to. The absence of significant pathology in the umbilical cords, along with the lack of association between certain placental pathologies and perinatal mortality and morbidity, have led both clinicians and pathologists to inadequately evaluate the placenta and umbilical cord. In our study, İnvestigators aimed to perform immunohistochemical and biochemical analysis by comparing two groups, one consisting of women who smoked throughout their pregnancy and the other of those who never smoked, including different markers in accordance with the literature.

Method: The pregnant women included in the study were categorized according to their smoking status as follows:

Group I: Non-smokers (smoking -) Group II: Smokers (smoking +) during pre-pregnancy and throughout the pregnancy In this study, 40 pregnant women who smoked during their pregnancy (between 37 and 42 weeks of gestation) and 37 age- and parity-matched healthy non-smoking pregnant women with full-term births between 37 and 42 weeks of gestation were selected as the control group. Umbilical cord samples (2 ml of blood and a 5 cm tissue sample) were collected from both groups without delay and fixed in 10% formalin. The tissue samples were processed for histological analysis with routine hematoxylin and eosin (H&E) staining following fixation in 10% formalin solution and routine paraffin embedding.

İnvestigators aimed to examine the presence of oncological factors such as CD44, CD34, CD90, and ALDH molecules in the umbilical cord tissue of smokers during pregnancy through immunohistochemistry, and to explore the biochemical relationship of these molecules with their counterparts, CD34, CD44, CD90, and ALDH, found in the umbilical cord blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnancy under 37 weeks
* Age range 18-50
* Being literate in Turkish
* Not having any additional disease
* Agreeing to participate in the study

Exclusion Criteria:

* High-risk pregnancies (gestational hypertension, preeclampsia, HELLP syndrome, chronic hypertension, gestational and pregestational diabetes, cholestasis, intrauterine growth retardation, etc.)
* Multiple pregnancy
* Pregnant women under the age of 18
* Smoking
* Medication use (excluding routinely used food supplements during pregnancy)
* Additional disease (thyroid, renal failure, liver failure, hepatitis, heart disease, connective tissue disease, etc.)
* Immunosuppressive use
* Presence of active or chronic infection
* Presence of active or chronic inflammatory disease
* Patients who gave birth at an external center or later chose to withdraw from the study
* Patients who did not have any exclusion criteria at the time of smokers or when blood was drawn for the control group, but who later developed any exclusion criteria.
* Premature birth of patients included in the control group

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women smokers pregnant women nonsmokers
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-01-14 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Hospitalized pregnant women's with smokers and nonsmokers 80%umblical cord tissues 3x3 cm collected while birth during the study .umblical tissues staining will be Measured by Cd34, Cd44, Cd90 and ALDH immunohistochemistry technique. | Baseline
Hospitalized pregnant women's with smokers and nonsmokers 80% umblical blood 5-7 ml collected while birth during the study. Bloods will be measured by Cd34, Cd44, Cd90 and ALDH biochemistry elisa technique. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hayrunnisa yeşil Sarsmaz, Manisa, Mani̇sa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided